CLINICAL TRIAL: NCT02609191
Title: Assessment of Body Composition Via Dual-energy X-ray Absorptiometry Bone Densitometry: Cross Calibration and Reproducibility Between the "Stratos DR" and "Discovery A" Bone Densitometers
Brief Title: Assessment of Body Composition Via Dual-energy X-ray Absorptiometry Bone Densitometry
Acronym: STRATOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: DMS Apelem (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LOCAL/2015/VB-01; 2015-A00987-42 (Other: ANSM)
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2017-10

CONDITIONS: Osteodensitometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The study population: first 30 patients (Experimental): The study population consists of adult patients referred to the Nuclear Medicine and Medical Biophysics Department of the Nîmes University Hospital for the performance of an osteodensitometric examination.
  Intervention: Whole body exam using the "Discovery A"
  Intervention: First whole body exam using the "Stratos DR"
  Intervention: Second whole body exam using the "Stratos DR"
  Interventions: Device: Whole body exam using the "Discovery A"; Device: First whole body exam using the "Stratos DR"; Device: Second whole body exam using the "Stratos DR"
- The study population: last 20 patients (Experimental): The study population consists of adult patients referred to the Nuclear Medicine and Medical Biophysics Department of the Nîmes University Hospital for the performance of an osteodensitometric examination.
  Intervention: Whole body exam using the "Discovery A"
  Intervention: First whole body exam using the "Stratos DR"
  Interventions: Device: Whole body exam using the "Discovery A"; Device: First whole body exam using the "Stratos DR"

INTERVENTIONS:
Device: Whole body exam using the "Discovery A" — Whole body exam using the "Discovery A" machine made by Hologic.
Device: First whole body exam using the "Stratos DR" — First whole body exam using the "Stratos DR" machine made by the DMS group.
Device: Second whole body exam using the "Stratos DR" — Second whole body exam using the "Stratos DR" machine made by the DMS group. This second exam is required for reproducibility purposes.
  Arms: The study population: first 30 patients

SUMMARY:
The main objective of this study is to validate the measurement characteristics of a new bone densitometer, the Stratos DR:

* Via cross calibration to the results of body composition (BC) measurement results to those of a reference device (the "Discover A" by Hologic) in terms of body fat percentage, lean mass percentage of total body mass and for different subregions (left and right arms, left and right sides, lumbar and thoracic spine, pelvis, left and right legs, head, android area, gynecoid area, visceral region).
* And by the evaluation of the reproducibility of the BC measurement results in terms of fat mass and lean mass.

DETAILED DESCRIPTION:
The secondary objective of this study is to cross calibrate the measures of bone mineral content (BMC) and bone mineral density (BMD) from the Stratos DR against those of the Discovery A on the whole body and its subregions.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is referred by a doctor for the performance of an osteodensitometry examination.

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection or any kind of guardianship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The subject is suffering from a visually significant scoliosis
* The patient is pregnant or breastfeeding
* Patient weighing over 160 kg
* Patient having undergone X-ray examination using a contrast medium such as barium in the 7 days preceding the visit
* Patient who underwent an examination using γ rays in the 15 days preceding the visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Lin concordance coefficient for fat mass | Day 0
  The cross calibration between the two devices (Stratos vs Discovery) in terms of fat mass and lean mass is estimated by the appreciation of the Lin concordance coefficient.
Lin concordance coefficient for lean mass | Day 0
  The cross calibration between the two devices (Stratos vs Discovery) in terms of fat mass and lean mass is estimated by the appreciation of the Lin concordance coefficient.
RMS-%CV (root-mean-square coefficient of variation) for total fat mass | Day 0
  Reproducibility will be evaluated in terms of RMS-% CV for calculating the value of the least significant change (LSC). The values of RMS-%CV (root-mean-square coefficient of variation) of the total fat mass and total lean mass will be compared with the limit values recommended by the ISCD. (International Society for Clinical Densitometry)
RMS-%CV (root-mean-square coefficient of variation) for total lean mass | Day 0
  Reproducibility will be evaluated in terms of RMS-% CV for calculating the value of the least significant change (LSC). The values of RMS-%CV (root-mean-square coefficient of variation) of the total fat mass and total lean mass will be compared with the limit values recommended by the ISCD. (International Society for Clinical Densitometry)

SECONDARY OUTCOMES:
Lin's concordance coefficient for Bone Mineral Content | Day 0
  The cross calibration between the two devices (Stratos vs Discovery) in terms of Bone Mineral Content and Bone Mineral Density will be estimated by the study of Lin's concordance coefficient.
Lin's concordance coefficient for Bone Mineral Density | Day 0
  The cross calibration between the two devices (Stratos vs Discovery) in terms of Bone Mineral Content and Bone Mineral Density will be estimated by the study of Lin's concordance coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Boudousq, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Neron M, Fatton B, Monforte M, Mares P, de Tayrac R, Letouzey V. [Evaluation of urine postvoid residuals in post-partum period: a prospective and descriptive clinical study]. Prog Urol. 2015 Mar;25(4):211-6. doi: 10.1016/j.purol.2014.09.043. Epub 2014 Oct 22. French. PMID 25450754